CLINICAL TRIAL: NCT00000885
Title: A Phase II Study of the Prolongation of Virologic Success (ACTG 372A) and Options for Virologic Failure (ACTG B/C/D) in HIV-Infected Subjects Receiving Indinavir in Combination With Nucleoside Analogs: A Rollover Study for ACTG 320
Brief Title: Treatment Success and Failure in HIV-Infected Subjects Receiving Indinavir in Combination With Nucleoside Analogs: A Rollover Study for ACTG 320
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 372; 11333 (Registry Identifier: DAIDS ES); ACTG 701; ACTG 702; ACTG 706
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Indinavir; RNA, Viral; Treatment Failure; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; abacavir; Nelfinavir; efavirenz; Carnitine; adefovir dipivoxil; Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Abacavir sulfate
Drug: Nelfinavir mesylate
Drug: Efavirenz
Drug: Levocarnitine
Drug: Adefovir dipivoxil
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
Group A:

To compare the time to confirmed virologic failure (2 consecutive plasma HIV-RNA concentrations of 500 copies/ml or more) between the treatment arms: abacavir (ABC) or placebo in combination with zidovudine (ZDV), lamivudine (3TC), and indinavir (IDV). To evaluate the safety and tolerability of these treatment arms. [AS PER AMENDMENT 06/16/99: To compare the time to confirmed treatment failure, permanent discontinuation of treatment, or death between the treatment arms.] [AS PER AMENDMENT 12/27/01: Groups B, C, and D completed follow-up on March 4, 1999. Therefore, only information pertinent to Group A is applicable.]

Group B:

To compare the proportion of patients who achieve plasma HIV-1 RNA concentrations below 500 copies/ml, as assessed by the standard Roche Amplicor assay at Week 16, or to compare the absolute changes in plasma HIV-1 RNA concentrations at Week 16 across the treatment arms: ABC or approved nucleoside analogs and nelfinavir (NFV) or placebo in combination with efavirenz (EFV) and adefovir dipivoxil. To compare the safety and tolerability of these treatment arms.

Group C:

To monitor plasma HIV-1 RNA trajectory over time and determine the time to a confirmed plasma HIV-1 RNA concentration above 2,000 copies/ml on 2 consecutive determinations for patients treated with ZDV or stavudine (d4T) plus 3TC and IDV.

Group D:

To evaluate plasma HIV-1 RNA responses at Weeks 16 and 48. To evaluate the safety and tolerability of the treatment arms: ABC, EFV, adefovir dipivoxil, and NFV.

This study explores new treatment options for ACTG 320 enrollees (and, if needed, a limited number of non-ACTG 320 volunteers) who have been receiving ZDV (or d4T) plus 3TC and IDV and are currently exhibiting a range of virologic responses. By dividing the study into the corresponding, nonsequential cohorts (Groups A, B, C, D), different approaches to evaluating virologic success, i.e., undetectable plasma HIV-1 RNA levels, and virologic failure, i.e., plasma HIV-1 RNA levels of 500 copies/ml or more [AS PER AMENDMENT 12/27/01: 200 copies/ml or more], are explored while maintaining long-term follow-up of ACTG 320 patients. [AS PER AMENDMENT 12/27/01: Groups B, C, and D completed follow-up on March 4, 1999. Therefore, only information pertinent to Group A is applicable. This study will examine the question of whether intensification of therapy can prolong the virologic benefit in individuals whose plasma HIV-1 RNA concentrations have been below the limits of assay detection on ZDV (or d4T) plus 3TC plus IDV.]

DETAILED DESCRIPTION:
This study explores new treatment options for ACTG 320 enrollees (and, if needed, a limited number of non-ACTG 320 volunteers) who have been receiving ZDV (or d4T) plus 3TC and IDV and are currently exhibiting a range of virologic responses. By dividing the study into the corresponding, nonsequential cohorts (Groups A, B, C, D), different approaches to evaluating virologic success, i.e., undetectable plasma HIV-1 RNA levels, and virologic failure, i.e., plasma HIV-1 RNA levels of 500 copies/ml or more [AS PER AMENDMENT 12/27/01: 200 copies/ml or more], are explored while maintaining long-term follow-up of ACTG 320 patients. [AS PER AMENDMENT 12/27/01: Groups B, C, and D completed follow-up on March 4, 1999. Therefore, only information pertinent to Group A is included. This study will examine the question of whether intensification of therapy can prolong the virologic benefit in individuals whose plasma HIV-1 RNA concentrations have been below the limits of assay detection on ZDV (or d4T) plus 3TC plus IDV.]

Rollover patients from ACTG 320 are given enrollment priority and permitted to enroll in all 4 study groups; non-ACTG patients are permitted to enroll in Groups A and B if accrual objectives are not met with ACTG 320 patients.

GROUP A:

Patients with screening plasma HIV-1 RNA concentrations below 500 copies/ml are randomized to 1 of 2 treatment arms and stratified according to their participation in ACTG 320 (original randomization to IDV versus open-label IDV). The 2 treatment arms are as follows:

ARM A1: IDV plus ZDV (or d4T) plus 3TC plus ABC. ARM A2: IDV plus ZDV (or d4T) plus 3TC plus ABC placebo. Patients who achieve a plasma HIV-1 RNA level of 500 copies/ml or more on 2 consecutive determinations may continue their assigned arm in a blinded fashion, or seek the best alternative therapy selected by the local investigator or primary care physician.

GROUP B:

Nonnucleoside reverse transcriptase inhibitor (NNRTI)-naive patients with plasma HIV-1 RNA plasma concentrations of 500 copies/ml or more are randomized to 1 of 4 treatment arms and stratified by plasma HIV-1 RNA concentrations (above versus below 15,000 RNA copies/ml) and participation in ACTG 320 (original randomization to IDV versus open-label IDV). The treatment arms are as follows:

ARM B1: ABC plus EFV plus adefovir dipivoxil plus NFV. ARM B2: ABC plus EFV plus adefovir dipivoxil plus NFV placebo. ARM B3: 2 nucleoside reverse transcriptase inhibitors (NRTIs) (or 1 if 2 not tolerated) (chosen from ZDV, 3TC, d4T, or didanosine [ddI]) plus EFV plus adefovir dipivoxil plus NFV.

ARM B4: 2 NRTIs (or 1 if 2 not tolerated) (chosen from ZDV, 3TC, d4T, or ddI) plus EFV plus adefovir dipivoxil plus NFV placebo.

GROUP C:

NNRTI-naive patients with plasma HIV-1 RNA concentrations of 500-2,000 copies/ml at screening may elect to be randomized to a treatment arm in Group B or continue with their current ACTG 320 regimen as follows:

ARM C: ZDV (or d4T) plus 3TC plus IDV. Patients who elect this treatment are randomized in Group B if their plasma HIV-1 RNA concentrations are confirmed to be above 2,000 copies.

GROUP D:

NNRTI-experienced, ACTG 320 patients with screening plasma HIV-1 RNA concentrations of 500 copies/ml or more receive open-label treatment as follows:

ARM D: ABC plus EFV plus adefovir dipivoxil plus NFV. [AS PER AMENDMENT 06/29/98: Enrollment to Group B is closed to accrual. Group A patients with HIV-1 RNA of 200 copies/ml or more on 2 consecutive determinations may continue their assigned treatment or seek best alternative antiretroviral therapy, which may include access to ABC. Group B patients with plasma HIV-1 RNA of 500 copies/ml or more may continue their assigned treatment or seek best available antiretroviral therapy, which may include access to ABC, EFV, and adefovir dipivoxil with L-carnitine supplementation. Group C patients with HIV-1 RNA levels above 2,000 copies/ml and Group D patients with levels above 500 copies/ml may no longer be randomized to a treatment arm in Group B. Such patients may continue their assigned treatment or seek best available therapy, which may include access to therapy as per Group B patients.] [AS PER AMENDMENT 06/16/99: Study treatment for Groups B, C, and D has been completed. Group A patients with a confirmed plasma HIV-2 endpoint who remain on study may have access to ABC while on study.] [AS PER AMENDMENT 12/27/01: With Version 4.0 of the protocol, many of the metabolic assessments and the cardiovascular risk assessment will be repeated, and a self-reported questionnaire of body shape changes will be added. In addition, an investigation of the effect of long-term IDV on pyuria/hematuria is added, as well as a study of HIV-1 RNA in peripheral blood mononuclear cells (PBMCs).]

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Chemoprophylaxis for Pneumocystis carinii pneumonia for all patients with a CD4 cell count of 200 cells/mm3 or less.

Allowed:

* Treatment, maintenance, or chemoprophylaxis, including topical and/or oral antifungal agents unless otherwise excluded by the protocol.
* All antibiotics as clinically indicated, unless otherwise excluded in the protocol.
* Systemic corticosteroid use for 21 days or less for acute problems as medically indicated. Chronic corticosteroid use is not permitted, unless it is within physiologic replacement levels. Study team must be contacted in these instances.
* rEPO and G-CSF as medically indicated.
* Regularly prescribed medications such as [AS PER AMENDMENT 06/29/98: alternative, FDA-approved antiretrovirals not supplied by the study] [AS PER AMENDMENT 12/27/01: or unapproved antiretrovirals available by expanded access (when permanently discontinued from randomized study treatment)], antipyretics, analgesics, allergy medications, antidepressants, sleep medications, oral contraceptives, megestrol acetate, testosterone, or any other medications not otherwise excluded by the protocol, as medically indicated.
* [AS PER AMENDMENT 12/27/01: Supplemental and] alternative therapies such as vitamins, acupuncture, and visualization techniques.

Recommended as an alternative agent for chemoprophylaxis against Mycobacterium avium complex for patients randomized to EFV in Group B or D:

* clarithromycin or azithromycin.

Patients must have:

* HIV-1 infection as documented by any licensed ELISA test kit and confirmed by either a Western Blot, HIV culture, HIV antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA at any time prior to study entry.

Non-ACTG patients:

* Documented CD4 cell count of 200 cells/mm3 or less at the time of initiation of ZDV (or d4T) plus 3TC plus IDV.
* Signed, informed consent from a parent or legal guardian for patients under 18 years of age.

Prior Medication:

Required:

Non-ACTG 320 patients:

* At least 3 months prior therapy with ZDV (or d4T) plus 3TC plus IDV and continued receipt of ZDV (or d4T) plus 3TC plus IDV until enrollment. IDV and 3TC must have been initiated concurrently.

ACTG patients:

* Randomization to the ZDV (or d4T) plus 3TC plus IDV combination arm or receipt of open-label prior to unblinding and maintenance of that treatment as participation in ACTG 320.

Group D:

* Prior NNRTI-exposure.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Unexplained temperature above 38.5 C for any 7 days or chronic diarrhea, defined as more than 3 liquid stools per day persisting for 15 days, within 30 days prior to study treatment.
* AIDS-related malignancy, other than minimal Kaposi's sarcoma that requires systemic chemotherapy. Minimal Kaposi's sarcoma is defined as 5 or fewer cutaneous lesions and no visceral disease or tumor-associated edema that does not require systemic therapy.
* Documented or suspected acute hepatitis within 30 days prior to study entry, irrespective of laboratory values.

Concurrent Medication:

Excluded:

* All antiretroviral therapies other than study [AS PER AMENDMENT 06/16/99: provided] medications, [AS PER AMENDMENT 06/16/99: unless approved by the protocol chairs] [AS PER AMENDMENT 12/27/01: while on original randomized treatment.]
* Rifabutin and rifampin.
* Investigational agents without specific approval from the protocol chair.
* Systemic cytotoxic chemotherapy.
* Oral ketoconazole and itraconazole. NOTE: Itraconazole may be permitted for Group B and Group D patients if fluconazole is not an option.
* Terfenadine, astemizole, cisapride, triazolam, midazolam, amiodarone, quinine, ergot derivatives, isotretinoin, [AS PER AMENDMENT 12/27/01: pimozide, St.John's Wort, and milk thistle.]
* [AS PER AMENDMENT 12/27/01: Concomitant use of lovastatin or simvastatin is not recommended because of potential drug interactions. Pravastatin or atorvastatin may be used after consultation with the Study Team.]

To be avoided:

* Herbal medications.

Prior Medication:

Excluded:

* Any prior protease inhibitor therapy other than indinavir.
* Interferons, interleukins, or HIV vaccines within 30 days prior to study entry.
* Any experimental therapy within 30 days prior to study entry.
* Rifampin, rifabutin, ketoconazole, or itraconazole within 14 days of study entry.

Non-ACTG patients:

* Acute therapy for an infection or other medical illness within 14 days prior to study therapy.
* NNRTI therapy prior to study entry (with the exception of Group D).
* Recombinant erythropoietin (rEPO), granulocyte colony-stimulating factor (G-CSF, filgrastim), or granulocyte-macrophage colony-stimulating factor (GM-CSF, sargramostim) within 30 days prior to study entry.

Caution should be taken in the consumption of alcoholic beverages with study medications.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440
Dates: Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hammer, Study Chair
Locations (53):
- United States (52):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Georgetown Univ Hosp, Washington D.C., District of Columbia
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - St Vincent's Hosp / Mem Sloan-Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Kentucky Lexington, Cincinnati, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas Galveston, Galveston, Texas
  - Univ Texas Health Science Ctr / Univ Texas Med School, Houston, Texas
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Henry K, Zackin R, Dube M, Hammer S, Currier J. ACTG 5056: metabolic status and cardiovascular disease risk for a cohort of HIV-1-infected persons durably suppressed on an indinavir-containing regimen (ACTG 372A). 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 656)
- [Background] Hammer S, Squires K, Degruttola V, Fischl M, Bassett R, Demeter L, Hertogs K, Larder B. Randomized trial of abacavir (ABC) & nelfinavir (NFV) in combination with efavirenz (EFV) & adefovir dipivoxil (ADV) as salvage therapy in patients with virologic failure receiving indinavir (IDV). Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:159 (abstract no 490)
- [Background] Hammer SM, Bassett R, Squires KE, Fischl MA, Demeter LM, Currier JS, Mellors JW, Morse GD, Eron JJ, Santana JL, DeGruttola V; ACTG 372B/D Study Team. A randomized trial of nelfinavir and abacavir in combination with efavirenz and adefovir dipivoxil in HIV-1-infected persons with virological failure receiving indinavir. Antivir Ther. 2003 Dec;8(6):507-18. No abstract available. PMID 14760884
- [Derived] Hammer SM, Ribaudo H, Bassett R, Mellors JW, Demeter LM, Coombs RW, Currier J, Morse GD, Gerber JG, Martinez AI, Spreen W, Fischl MA, Squires KE; AIDS Clinical Trials Group (ACTG) 372A Study Team. A randomized, placebo-controlled trial of abacavir intensification in HIV-1-infected adults with virologic suppression on a protease inhibitor-containing regimen. HIV Clin Trials. 2010 Nov-Dec;11(6):312-24. doi: 10.1310/hct1106-312. PMID 21239359